CLINICAL TRIAL: NCT07382024
Title: Efficacy of Tirzepatide on Weight Loss and Atrial Fibrillation Burden After Catheter Ablation in Overweight or Obese Patients
Brief Title: Tirzepatide to Reduce rEcurrence And Burden After Ablation of Atrial Fibrillation
Acronym: TREAT-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending Physician, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Temporary number -29569
Record Dates: First submitted 2026-01-08; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation Ablation; Persistent Atrial Fibrillation; Obesity & Overweight
Keywords: Atrial fibrillation; Catheter ablation; Tirzepatide; Overweight and obesity; AF burden; Recurrence; Quality of life
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Overweight; Recurrence | interventions — Tirzepatide; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, parallel-group randomized controlled trial. Eligible patients with persistent atrial fibrillation scheduled for de novo catheter ablation are randomized in a 1:1 ratio to receive tirzepatide plus standard peri-procedural and post-ablation care or standard care alone. Participants remain in their originally assigned treatment group for all analyses according to the intention-to-treat principle.
Masking Description: Although participants and treating investigators are not masked to treatment assignment (open-label design), the independent Endpoint Assessment Committee is fully blinded to group allocation when adjudicating the primary endpoint of atrial fibrillation burden and other adjudicated outcomes, using de-identified ECG and clinical data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care（Intervention: Other - standard care / no tirzepatide） (Active Comparator)
  Interventions: Other: Standard Care (in control arm)
- Tirzepatide + Standard Care（Intervention: Drug - tirzepatide） (Active Comparator)
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Subcutaneous tirzepatide 2.5 mg once weekly, initiated approximately 4 weeks before the scheduled de novo catheter ablation and continued for 3 months after the procedure (total treatment duration about 4 months), in addition to standard peri-procedural and post-ablation care.
  Arms: Tirzepatide + Standard Care（Intervention: Drug - tirzepatide）
Other: Standard Care (in control arm) — Standard peri-procedural and post-ablation care for persistent atrial fibrillation without tirzepatide or other study-specific metabolic pharmacotherapy.
  Arms: Standard Care（Intervention: Other - standard care / no tirzepatide）

SUMMARY:
The goal of this clinical trial is to determine whether tirzepatide can reduce atrial fibrillation (AF) burden after catheter ablation in overweight or obese patients with persistent AF. It will also evaluate the effects of tirzepatide on body weight, metabolic risk factors, and clinical outcomes, as well as its safety and tolerability in this population.

The main questions it aims to answer are:

1. Does peri-procedural treatment with tirzepatide reduce AF burden at 3 months after de novo catheter ablation, as measured by 7-day continuous ECG patch monitoring?
2. Does tirzepatide lead to greater weight loss and improvement in metabolic parameters compared with standard care alone?
3. Does tirzepatide reduce AF recurrence and cardiovascular events during 12 months of follow-up? Researchers will conduct a multi-center, open-label, endpoint-blinded, randomized controlled trial in adults aged 18-80 years with persistent AF and body mass index ≥25 kg/m² who are scheduled for de novo catheter ablation. Participants will be randomized 1:1 to receive either tirzepatide plus standard peri-procedural and post-ablation care or standard care alone.

Participants in the tirzepatide group will receive subcutaneous tirzepatide 2.5 mg once weekly starting about 4 weeks before ablation and continuing for 3 months afterward, for a total treatment duration of approximately 4 months. All participants will be followed at 1, 2, 3, 6, and 12 months after ablation, with detailed assessment of AF burden, AF recurrence, echocardiographic parameters, metabolic profile, quality of life by the AFEQT questionnaire, and safety events.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common sustained arrhythmias and is associated with increased risks of stroke, heart failure, cognitive decline, and mortality, creating a substantial burden for patients and healthcare systems. Catheter ablation has become an important rhythm-control strategy that can restore sinus rhythm and improve quality of life in patients with AF. However, 30-50% of patients still experience recurrent atrial tachyarrhythmias after ablation, and higher AF burden has been linked to worse clinical outcomes, making AF burden a clinically relevant endpoint beyond a simple yes/no definition of recurrence.

Obesity and metabolic dysfunction are major upstream drivers of AF, promoting atrial structural and electrical remodeling through hemodynamic load, epicardial fat accumulation, systemic inflammation, and neurohormonal activation. Intensive lifestyle and risk-factor management programs can reduce AF burden and improve ablation outcomes, but such interventions are often difficult to implement and sustain in routine practice. Pharmacologic therapies that induce substantial and durable weight loss and improve cardiometabolic risk may therefore offer a practical strategy to lower AF burden after ablation in overweight or obese patients.

Tirzepatide is a dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 (GLP-1) receptor agonist that has produced large and sustained weight loss and broad cardiometabolic benefits in patients with obesity and type 2 diabetes, including improvements in glycemic control, blood pressure, and lipid profiles. In high-risk cardiometabolic populations, tirzepatide has also been associated with reductions in heart failure events and markers of congestion, suggesting favorable effects on cardiac loading conditions and structural remodeling. These data provide a strong rationale to test whether tirzepatide-induced weight loss and metabolic improvement can translate into reduced AF burden after catheter ablation.

The TREAT-AF trial is an investigator-initiated, multi-center, open-label, endpoint-blinded randomized controlled trial in adults with persistent AF and body mass index ≥25 kg/m² who are scheduled for de novo catheter ablation. Participants are randomized 1:1 to receive peri-procedural tirzepatide in addition to standard care or standard care alone. Tirzepatide is started approximately 4 weeks before the ablation procedure and continued for 3 months afterward, aligning pharmacologic weight loss and metabolic optimization with the period of atrial healing and electrical remodeling after ablation. AF burden at 3 months is assessed by 7-day single-lead ECG patches and adjudicated by a blinded endpoint assessment committee. Secondary assessments include AF recurrence, echocardiographic measures of left atrial structure, metabolic parameters, quality of life using the AFEQT questionnaire, and cardiovascular events through 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Diagnosed with persistent atrial fibrillation and scheduled for de novo catheter ablation.
3. Body mass index (BMI) ≥ 25 kg/m² at screening.
4. Able and willing to provide written informed consent.

Exclusion Criteria:

1. Long-standing AF or marked left atrial enlargement (persistent AF duration > 5 years or left atrial anterior-posterior diameter > 50 mm).
2. AF secondary to reversible causes (e.g., hyperthyroidism, acute infection, acute pulmonary embolism, recent cardiac surgery).
3. Severe structural heart disease that may significantly affect ablation outcomes (e.g., hypertrophic cardiomyopathy, rheumatic valvular disease, dilated cardiomyopathy).
4. Planned major non-AF-related surgery or interventional procedure within 3 months.
5. Other arrhythmias requiring chronic antiarrhythmic drug therapy.
6. Intracardiac thrombus or any contraindication to catheter ablation as judged by the investigator.
7. Active systemic infection at screening.
8. Contraindications to tirzepatide or GLP-1/GIP receptor agonists (e.g., prior serious hypersensitivity, personal or family history of medullary thyroid carcinoma or MEN2, history of clinically significant pancreatitis, severe gastrointestinal disease that may impair tolerance or absorption).
9. Poorly controlled type 1 diabetes, recent diabetic ketoacidosis, end-stage renal disease requiring dialysis, or severe hepatic dysfunction judged clinically significant.
10. Pregnancy, breastfeeding, or women of childbearing potential unwilling or unable to use adequate contraception during the study.
11. Participation in another interventional clinical study within 30 days prior to screening or planned participation during the study period.
12. Any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation, including inability to comply with study procedures or follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden at 3 months after catheter ablation | 3 months after catheter ablation (7-day ECG patch monitoring period)
  AF burden is defined as the proportion of time an individual is in any atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) during a 7-day monitoring period, assessed using continuous single-lead ECG patch recordings. AF burden will be adjudicated by a blinded Endpoint Assessment Committee based on de-identified ECG data.

SECONDARY OUTCOMES:
Atrial fibrillation recurrence within 3 months after catheter ablation | From the date of ablation to 3 months after ablation
  AF recurrence is defined as the first documented episode of any atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) lasting ≥30 seconds, detected by ECG monitoring or clinically indicated ECG during the first 3 months after ablation. Episodes occurring within a standard blanking period, if applicable, will be handled according to the study protocol.
Change in left atrial structure by echocardiography at 3 months | Baseline and 3 months after ablation
  Change from baseline to 3 months in echocardiographic measures of left atrial structure (left atrial volume indices), assessed by transthoracic echocardiography according to standard guidelines.
Change in atrial fibrillation-related quality of life (AFEQT score) | Baseline and 3 months after ablation
  Change from baseline to 3 months in health-related quality of life as measured by the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire, using a validated Chinese version for Chinese-speaking participants. Higher scores indicate better quality of life.
Atrial fibrillation recurrence within 12 months after catheter ablation | From the date of ablation to 12 months after ablation
  Time to first recurrence of any atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) lasting ≥30 seconds, detected by ECG or rhythm monitoring during 12 months of follow-up after ablation.
Cardiovascular death or cardiovascular hospitalization within 12 months | From the date of ablation to 12 months after ablation
  Composite of cardiovascular death or hospitalization for cardiovascular causes (e.g., heart failure, acute coronary syndrome, stroke, or other predefined cardiovascular events), defined according to consensus cardiovascular endpoint definitions and adjudicated by the Endpoint Assessment Committee.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Cardiovascular Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not planned at this time because the protocol and consent forms were not specifically designed for external data sharing. Future sharing may be reconsidered if appropriate regulatory approvals, institutional policies, and participant consent can be ensured.